CLINICAL TRIAL: NCT01072617
Title: Safety and Therapeutic Efficacy of Cerebellar Repetitive Transcranial Magnetic Stimulation in Patients With Schizophrenia
Brief Title: Cerebellar rTMS for the Treatment of Schizophrenic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Alvaro Pascual-Leone, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007P000395
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety of rTMS in schizophrenia patients (Experimental): Participants will receive repetitive transcranial magnetic stimulation via MagPro x100 device to the vermis of cerebellum twice a day over 5 days
  Interventions: Device: Transcranial magnetic stimulation via MagPro x100 device

INTERVENTIONS:
Device: Transcranial magnetic stimulation via MagPro x100 device — Participants will receive 10 repetitive transcranial magnetic stimulation sessions to the vermis of cerebellum using the MagPro x100 TMS device. These 10 rTMS sessions will be administered from Monday to Friday in five days, twice a day with a minimum of 4-hour gap between the sessions. Repetitive TMS will be applied with the intermittent theta burst pattern (iTBS). These parameters are known to cause excitation in brain activity.
  Anatomically precise localization of rTMS will be achieved using a frameless stereotactic system.

SUMMARY:
The primary aim of this protocol is to determine whether the use of repetitive transcranial magnetic stimulation (rTMS) over vermis of the cerebellum may be safe and therapeutically effective in patients with schizophrenia. Because this is the first evaluation of this treatment in this population, the focus of this study is safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years
2. Diagnosis of schizophrenia according to DSM-IV criteria(by a board-certified psychiatrist)

Exclusion Criteria:

1. Prior neurosurgical procedures
2. Any history of seizure
3. Previous head injury
4. Contraindication to TMS:

   1. Implanted pacemaker
   2. Medication pump
   3. Vagal stimulator
   4. Deep brain stimulator
   5. Metallic hardware in the head or scalp: shrapnel, surgical clips, or fragments from welding
   6. Signs of increased intracranial pressure
5. TENS unit and ventriculo-peritoneal shunt
6. Pregnancy or lactating; note that a negative pregnancy test will be required if the patient is a female in reproductive years
7. Advanced liver, kidney, cardiac, or pulmonary disease as defined clinically or a terminal medical diagnosis consistent with survival < 1 year
8. A history of significant alcohol or drug abuse in the prior six months
9. No focal cortical insult can be present, including tumor or vascular malformation
10. Patients may not be actively enrolled in a separate intervention study
11. Patients unable to undergo a brain MR:

    a. claustrophobia refractory to anxiolytics ferromagnetic metal in the body such as a prosthetic heart valve, a pacemaker, or a brain aneurysm clip).
12. Change in antipsychotic medication during the last 4 weeks
13. Any emergency psychiatry department visit during the last 4 weeks
14. Been an inpatient in a psychiatry clinic within the last month
15. Any other axis I diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pascual-Leone, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety of rTMS in Schizophrenia Patients: Participants will receive repetitive transcranial magnetic stimulation via MagPro x100 device to the vermis of cerebellum twice a day over 5 days
  Transcranial magnetic stimulation via MagPro x100 device: Participants will receive 10 repetitive transcranial magnetic stimulation sessions to the vermis of cerebellum using the MagPro x100 TMS device. These 10 rTMS sessions will be administered from Monday to Friday in five days, twice a day with a minimum of 4-hour gap between the sessions. Repetitive TMS will be applied with the intermittent theta burst pattern (iTBS). These parameters are known to cause excitation in brain activity.
  Anatomically precise localization of rTMS will be achieved using a frameless stereotactic system.
Period: Overall Study
Arm/Group | Safety of rTMS in Schizophrenia Patients
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Safety of rTMS in Schizophrenia Patients
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Adverse event collection at baseline, daily for 5 days during treatment, every other day by phone until the final assessment at week 1 follow up visit.
Time Frame: 3 weeks
Measure: Number; unit: event
Arm/Group | Safety of rTMS in Schizophrenia Patients
Number analyzed (Participants) | 8
event | 1

2. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) - Positive Subscale
Description: Potential therapeutic efficacy was evaluated with the Positive and Negative Syndrome Scale (PANSS) Positive Subscale, a 7 item subscale measuring the presence/absence and severity of positive symptoms of schizophrenia. The minimum score is 7 and the maximum score is 49, with higher values representing greater symptom severity. Therapeutic efficacy was assessed at baseline, after 5 days of treatment, and 1 week post treatment. The overall PANSS total score (minimum = 30, maximum = 210) is computed by summing the positive, negative, and general subscales; and higher values represent more severe schizophrenia psychopathology.
Time Frame: Baseline, 5 days (post-treatment), 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Safety of rTMS in Schizophrenia Patients
Number analyzed (Participants) | 8
percentage of change
  Before treatment (baseline) | 17.13 (5.69)
  Last day of treatment (after 5 days of treatment) | 17 (5.93)
  1 week post treatment follow-up | 16.25 (5.12)

3. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) - Negative Subscale
Description: Potential therapeutic efficacy was evaluated with the Positive and Negative Syndrome Scale (PANSS) Negative Subscale, a 7 item subscale measuring the presence/absence and severity of negative symptoms of schizophrenia. The minimum score is 7 and the maximum score is 49, with higher values representing greater symptom severity. Therapeutic efficacy was assessed at baseline, after 5 days of treatment, and 1 week post treatment. The overall PANSS total score (minimum = 30, maximum = 210) is computed by summing the positive, negative, and general subscales; and higher values represent more severe schizophrenia psychopathology.
Time Frame: Baseline, 5 days (post-treatment), 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Safety of rTMS in Schizophrenia Patients
Number analyzed (Participants) | 8
percentage of change
  Before treatment (baseline) | 23.75 (6.92)
  Last day of treatment (after 5 days of treatment) | 19.75 (4.3)
  1 week post treatment follow-up | 19.88 (5.82)

4. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) - General Subscale
Description: Potential therapeutic efficacy was evaluated with the Positive and Negative Syndrome Scale (PANSS) General Subscale, a 16 item subscale measuring the presence/absence and severity of general psychopathology of schizophrenia. The minimum score is 16 and the maximum score is 112, with higher values representing greater psychopathology severity. Therapeutic efficacy was assessed at baseline, after 5 days of treatment, and 1 week post treatment. The overall PANSS total score (minimum = 30, maximum = 210) is computed by summing the positive, negative, and general subscales; and higher values represent more severe schizophrenia psychopathology.
Time Frame: Baseline, 5 days (post-treatment), 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Safety of rTMS in Schizophrenia Patients
Number analyzed (Participants) | 8
percentage of change
  Before treatment (baseline) | 41.38 (10.84)
  Last day of treatment (after 5 days of treatment) | 39.13 (11.81)
  1 week post treatment follow-up | 37 (9.1)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Safety of rTMS in Schizophrenia Patients
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety of rTMS in Schizophrenia Patients (N=8)
High blood pressure (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No